CLINICAL TRIAL: NCT01594099
Title: Weekly Cisplatin or Weekly Liposome Paclitaxel Concurrent Radiation Therapy in Treating Elderly People With Cervical Cancer
Brief Title: Concurrent Chemoradiotherapy for Cervical Cancer in Elderly Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Liu Zi, Profesor, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCR-02
Record Dates: First submitted 2012-03-27; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; elderly women; concurrent chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Radiotherapy alone (Active Comparator)
  Interventions: Radiation: irradiation
- Radiotherapy plus cisplatin (Experimental)
  Interventions: Drug: Cisplatin
- Radiotherapy plus liposome paclitaxel (Experimental)
  Interventions: Drug: liposome paclitaxel

INTERVENTIONS:
Radiation: irradiation — EBRT: 3D-CRT pelvic radiation, 95%CTV DT 50.4Gy/28f. Radiation volume Cover the gross disease, whole uterus ,parametria, and regional lymph nodes area. Upper border：branching of abdominal aorta. Lower border: the inferior margin of obturator foramen.
  Brachytherapy :Using an intrauterine tandem and colpostats. The total dose of A point is DT 20-25Gy/4-5f (EQD2=25-31.25 Gy，α/β=10).
  Other Names: RT
  Arms: Radiotherapy alone
Drug: Cisplatin — EBRT: 3D-CRT pelvic radiation, 95%CTV DT 50.4Gy/28f. Radiation volume Cover the gross disease, whole uterus ,parametria, and regional lymph nodes area. Upper border：branching of abdominal aorta. Lower border: the inferior margin of obturator foramen.
  Brachytherapy: Using an intrauterine tandem and colpostats. The total dose of A point is DT 20-25Gy/4-5f (EQD2=25-31.25 Gy，α/β=10).
  Chemotherapy: Cisplatin (20mg /week) will be carry out in the 2nd to 6th week during radiation therapy.
  Other Names: RT+C
  Arms: Radiotherapy plus cisplatin
Drug: liposome paclitaxel — EBRT: 3D-CRT pelvic radiation, 95%CTV DT 50.4Gy/28f. Radiation volume Cover the gross disease, whole uterus ,parametria, and regional lymph nodes area. Upper border：branching of abdominal aorta. Lower border: the inferior margin of obturator foramen.
  Brachytherapy: Using an intrauterine tandem and colpostats. The total dose of A point is DT 20-25Gy/4-5f (EQD2=25-31.25 Gy，α/β=10).
  Chemotherapy: Liposome paclitaxel (40mg /m2/2weeks) will be carry out in the 2nd ,4th,6th week during radiation therapy.
  Other Names: RT+Lp
  Arms: Radiotherapy plus liposome paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficiency and safety of weekly Cisplatin /Liposome paclitaxel concurrent chemoradiothrapy in the treatment of locally advanced cervical cancer in elderly women.

DETAILED DESCRIPTION:
Concurrent radiotherapy is the standard treatment of inoperable cervical cancer .Due to the physical conditions, elderly patients usually associated with medical complications, so generally just receive radiotherapy alone. Recently, some retrospective studies have shown that the impact of chemotherapy did not cause an increase in the complication rate among elderly patients as compared to younger patients with cervical cancer, and may improve the survival when concurrent with radiotherapy. Cisplatin and paclitaxel are two effective drug in treating cervical cancer, but whether they are safe enough for elderly when concurrent with radiotherapy, there are no clearly reports. In this study ,we replace the conventional dose chemotherapy with weekly cisplatin or lipsome paclitaxel , to compare the efficiency and safety of weekly cisplatin / liposome paclitaxel concurrent chemoradiotherapy and radiotherapy alone in the treatment of cervical cancer in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven squamous carcinoma of cervix
2. FIGO stageⅡB and ⅢB
3. Over 65 years
4. Do not receive other treatment
5. Performance index ECOG grade 0 to 2
6. Normal ECG
7. Normal hematological parameters
8. Normal renal and liver function tests

Exclusion Criteria:

1. Concomitant disease which may adversely affect the outcome
2. Poor nutritional status
3. Medical or psychological condition precluding treatment
4. Previous treatment
5. Concurrent treatment for any cancer

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-10 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1 month after the treatment completed
  Objective Response Rate: Complete response (CR)+ Partial response (PR) rates base on RECIST evaluation system.
Adverse Events | Participants will be followed from the treatment begin to 1 month after the treatment end.
  Record the Number of participants with adverse events and the Grades of the AE according to CTCAE v3.0

SECONDARY OUTCOMES:
Local Control Rate | Participants will be followed every year for the duration of 5 years
Tumor Free Survival Rate | From date of randomization until tumor recurrence or metastasis,assessed up to 5 years
Overall Survival Rate | From date of randomization until the date of death from any cause,assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Chen M W, M.D, Study Director — Affiliated Hospital of Medical College of Xi'an Jiaotong University